CLINICAL TRIAL: NCT05362266
Title: Incidence and Risk Factors of in Hospital Adverse Events in Acute Limb Ischemic Patient Undergoing Revascularization Treatment: a Retrospective Cohort Study
Brief Title: Adverse Events in Acute Limb Ischemic Patient Undergoing Revascularization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 052/2565
Record Dates: First submitted 2022-04-11; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Major Adverse Cardiac Events; Adverse Effect of Unspecified General Anesthetic
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute limb ischemia is one of the devastating vascular emergencies that lead to life and limb loss if the appropriate treatment is not reached.The revascularization is a cornerstone in treating acute limb ischemia. The conventional surgical approach includes surgical embolectomy and surgical bypass.From the anesthetic aspect, this emergency condition limits the lengthening cardiovascular assessment of this high-risk patient group which might lead to the uncertainty outcome.With the variety of patients and procedures, we sought to find out the perioperative adverse events, especially major adverse cardiac events, in acute ischemic limb patients undergoing revascularization, in order to increase awareness of the team and properly admit to ICU in a retrospective manner.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years
* undergoing revascularization surgery or procedure (surgical revascularization, endovascular revascularization, hybrid revascularization, catheter directed thrombolysis)

Exclusion Criteria:

* incomplete data during perioperative period

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age more than 18, with acute limb ischemia undergoing revascularization procedure
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiac events | during hospital stay, up to 4 weeks
  Incidence of major adverse cardiac events, which are cardiovascular death, myocardial infarction, stroke

SECONDARY OUTCOMES:
Incidence of the perioperative complication | during hospital stay, up to 4 weeks
  Incidence of the perioperative other complication, which are major bleeding, repercussion syndrome, compartment syndrome, rhabdomyolysis and unplanned ICU admission from any causes.
Factors contribute to the adverse outcome | during hospital stay, up to 4 weeks
  Factors contribute to the adverse outcome, which are the patients' condition and the underlying diseases, the surgical intervention and the anesthetic technique.

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Anesthesiology department, Siriraj Hospital, Mahidol University, Bangkok
  - MahidolU, Bangkok

IPD SHARING:
Plan to Share IPD: No
The data has no plan for sharing.